CLINICAL TRIAL: NCT01541137
Title: NSAID With IV-PCA Morphine is an Alternative to Thoracic Epidural Analgesia in Post-thoracotomy Pain
Brief Title: NSAIDs With Morphine-PCA Compared to Epidural Analgesia in Thoracotomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Academy of Finland (Other)
Responsible Party: Principal Investigator, Elina Tiippana, MD, M.D., Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 74555
Record Dates: First submitted 2012-02-18; First posted 2012-02-29 (Estimated); Last update posted 2012-02-29 (Estimated); Status verified 2012-02

CONDITIONS: Postoperative Pain
Keywords: thoracotomy; pain; NSAID; PCA; TEA; chronic
MeSH Terms: conditions — Pain, Postoperative; Pain; Bronchiolitis Obliterans Syndrome | interventions — Diclofenac; parecoxib; valdecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- diclofenac + IV-PCA (Active Comparator): oral diclofenac 75 mg, a 44-hour iv-infusion of diclofenac 150 mg/24h, intercostal nerve block with 20 ml of 0.5% bupivacaine, IV-PCA programmed with morphine boluses, from the 2nd postoperative morning the patients were given oral diclofenac 75 mg x 2, IV-PCA-morphine was discontinued after removal of pleural drains, and the patients were given oral oxycodone
  Interventions: Drug: Diclofenac
- parecoxib/ valdecoxib + IV-PCA (Active Comparator): oral valdecoxib 40 mg, a 44-hour iv-infusion parecoxib 80 mg/24h, intercostal nerve block with 20 ml of 0.5% bupivacaine, IV-PCA programmed with morphine, From the 2nd postoperative morning valdecoxib 40 mg x 2, IV-PCA-morphine was discontinued after removal of pleural drains, and the patients were given oral oxycodone
  Interventions: Drug: parecoxib/ valdecoxib
- patient controlled epidural analgesia (Active Comparator): At the induction of anesthesia the PCEA-patients were given IV paracetamol 1g and an epidural loading dose of 1 ml/10 kg of 0.15% bupivacaine with fentanyl 6 µg/ml. Thereafter a continuous infusion was started at 1 ml/10 kg/h. In the PACU PCEA-patients could take incremental doses, IV paracetamol 1g x 4 for the first 24 hours and thereafter 1g x 3 orally, PCEA was discontinued and paracetamol was replaced with ibuprofen 600 mg x 3 and oral oxycodone
  Interventions: Device: patient controlled epidural analgesia

INTERVENTIONS:
Drug: Diclofenac — oral diclofenac 75 mg, a 44-hour iv-infusion of diclofenac 150 mg/24h, oral diclofenac 75 mg x 2, IV-PCA programmed with morphine boluses of 2-3 mg and a lock-out time of 5-15 minutes
  Arms: diclofenac + IV-PCA
Drug: parecoxib/ valdecoxib — oral valdecoxib 40 mg, a 44-hour iv-infusion of parecoxib 80 mg/24h, IV-PCA programmed with morphine boluses of 2-3 mg and a lock-out time of 5-15 minutes
  Arms: parecoxib/ valdecoxib + IV-PCA
Device: patient controlled epidural analgesia — epidural catheter, epidural loading dose of 1 ml/10 kg of 0.15% bupivacaine with fentanyl 6 µg/ml. Thereafter a continuous infusion was started at 1 ml/10 kg/h. In the PACU PCEA-patients could take incremental doses of 3 ml with a 8-15 min lock-out time
  Arms: patient controlled epidural analgesia

SUMMARY:
The investigators investigated whether a strictly controlled pain management with patients participating in a clinical study can attenuate persistence of post-thoracotomy pain. The investigators also wanted to find out whether NSAID + intravenous patient-controlled analgesia with morphine is an efficacious alternative to thoracic epidural analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective thoracotomy for lung surgery

Exclusion Criteria:

* Contraindication to any of the study drugs or an epidural catheter,
* Significant liver, renal or cardiac disease
* Peptic ulcer
* Regular use of analgesics
* Re-thoracotomy, and the patient´s inability to understand the use of PCA/patient controlled thoracic epidural analgesia (PCEA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-03; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
pain intensity 6 months after surgery | 6 months
  The primary outcome when comparing the Intervention and Control groups was pain intensity 6 months after surgery.

SECONDARY OUTCOMES:
consumption of PCA-morphine | 4 days
  consumption of PCA-morphine in groups 1 and 2
pain intensity while coughing | 4 days
  pain intensity while coughing during the first four postoperative days using VAS (visual analogue scale) 0-10 cm (0 = no pain and 10 = worst imaginable pain) or NRS in the PACU (numeric rating scale, 0-10)
adverse effects | 1-7 days
  adverse effects (e.g. nausea, itching, sedation and subjective tiredness) measured with VAS 0-10 cm

CONTACTS AND LOCATIONS:
Overall Officials: Elina Tiippana, M.D., Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland